CLINICAL TRIAL: NCT05805761
Title: Antimicrobial Photodynamic Therapy With Erythrosine and Blue Light on Dental Biofilm Bacteria - Study Protocol for Randomized Clinical Trial
Brief Title: Antimicrobial Photodynamic Therapy With Erythrosine and Blue Light on Dental Biofilm Bacteria
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Marcela Leticia Leal Gonçalves, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EritroBiofilm
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment Group (Experimental): Participants in this group will receive the conventional treatment for the removal of dental biofilm (prophylaxis with bicarbonate jet).
  Interventions: Procedure: Conventional Treatment
- aPDT + Conventional Treatment Group (Experimental): Participants in this group will receive both the antimicrobial photodynamic therapy and the conventional treatment (prophylaxis with bicarbonate jet) for the removal of dental biofilm.
  Interventions: Procedure: Conventional Treatment; Procedure: Antimicrobial Photodynamic Therapy

INTERVENTIONS:
Procedure: Conventional Treatment — A bicarbonate jet will be used to remove the biofilm from the surface of the teeth.
Procedure: Antimicrobial Photodynamic Therapy — aPDT will be performed before each cleaning/prophylaxis session, only in one of the groups. Participants will swish with the photosensitizer erythrosine for 1 min of pre-irradiation time, so that the drug can stain all the bacterial biofilm. The D-2000 LED (DMC) will be applied, emitting at a wavelength of ʎ = 430-490 nm and 900-1100 mW/cm2. Irradiation will be performed until the biofilm of the cervical region is illuminated for 2 min per point. Each irradiation point will be approximately 0.4 cm2.
  Arms: aPDT + Conventional Treatment Group

SUMMARY:
The objective of this study is to investigate the effect of Antimicrobial Photodynamic Therapy mediated by Erythrosine and blue LED in the reduction of bacteria in dental biofilm. This clinical trial will be carried out with 30 patients who have biofilm, but without the presence of periodontal pockets, and who are being treated at the Dental Clinic of Universidade Metropolitana de Santos. A split-mouth model will be used (n = 30), with group I control - conventional treatment and group II - conventional treatment and antimicrobial photodynamic therapy (aPDT). The bicarbonate jet will be used to remove dental biofilm in both groups. The treatment will be carried out in 1 session. aPDT will be performed before cleaning/prophylaxis, only in group II. Participants will rinse with the photosensitizer erythrosine (diluted to 1mM) for 1 min of pre-irradiation time, so that the drug can stain all the bacterial biofilm. Then, the D-2000 LED (DMC) will be applied, emitting at a wavelength of ʎ = 430-490 nm and 900-1100 mW/cm2. Irradiation will be performed until the biofilm of the cervical region is illuminated for 2 min per point. Each irradiation point will be approximately 0.4 cm2. The microbiological examination will be performed from samples of supragingival biofilm collected from the gingival sulcus. Two collections will be performed in each experimental site before irradiation, and immediately after the irradiation procedure (group II) or prophylaxis (groups I and II). Biofilm samples will be collected before and after exposure, respectively, and sent to the microbiological laboratory for colony counting. After this period, the CFU's will be counted and the data will be submitted to statistical analysis for comparison of pre and post-treatment results and between groups (conventional X aPDT).

ELIGIBILITY:
Inclusion Criteria:

* The participant must present between 25% and 50% of biofilm index;
* Have at least 20 teeth present, without clinical probing depths greater than 3 mm.

Exclusion Criteria:

* Smokers;
* Uncontrolled diabetics or hypertensives;
* Cancer or its treatment;
* Pregnant women;
* Use of antibiotics in the last 6 months;
* Coagulation disorders (use of anticoagulants, presence of liver diseases, thrombocytopenia and immunosuppression);
* Patients undergoing orthodontic treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Colony Forming Units | Baseline and immediately after treatment.
  The microbiological examination will be carried out from biofilm samples collected from the gingival sulcus. Two collections will be performed in each experimental site before irradiation, and immediately after the prophylaxis procedure or irradiation. To collect the subgingival biofilm, the teeth will be isolated with cotton rolls, the supragingival biofilm will be removed with sterile gauze, and the subgingival biofilm sample will be obtained by introducing a tip of sterile absorbent paper (#30) inside of the periodontal pocket, being kept in position for 30 s. The tips will be removed and stored in properly identified sterile plastic microtubes, each tube containing 1 mL of sterile Brain Heart Infusion (BHI) culture medium will be packed on ice and analyzed immediately after collection.
  The samples will be used to determine the CFU's (Colony Forming Units). Each tube with 1 mL BHI will be vortexed and will undergo serial dilution from 10-1 to 10-5 times the original concentration.

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated in the study will be available from the corresponding author at a reasonable request. Once the data is entered electronically, participants identification details will no longer be attached to their data, they will be reported only by numbers. After the analysis of the data, volunteers will be invited to a meeting and the results will be shared, in case they wish to attend it. The authors intend to publish the results in a peer-review jornal and present them in cientific events.

REFERENCES:
- [Derived] Goncalves MLL, Sobral APT, Gallo JMAS, Gimenez T, Ferri EP, Ianello S, Motta PB, Motta LJ, Horliana ACRT, Santos EM, Bussadori SK. Antimicrobial photodynamic therapy with erythrosine and blue light on dental biofilm bacteria: study protocol for randomised clinical trial. BMJ Open. 2023 Sep 19;13(9):e075084. doi: 10.1136/bmjopen-2023-075084. PMID 37730405